CLINICAL TRIAL: NCT01890512
Title: INGENIO MRI/ FINELINE II ImageReadyTM Pacing System Data Collection in Patients Undergoing Magnetic Resonance Imaging
Brief Title: INGENIO MRI/ FINELINE II Pacing System Data Collection in Patients Undergoing MRI
Acronym: INFINITE-MRI
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C1897
Record Dates: First submitted 2013-06-25; First posted 2013-07-01 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2014-05

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ImageReady Pacemaker: patients previously implanted with a Boston Scientific MR Conditional pacemaker(ImageReady)

SUMMARY:
The INFINITE MRI Study is a prospective, non-randomized, multicenter, single arm study aimed at collecting data on ImageReady™ MR Conditional Pacing System (consisting of an INGENIO™ MRI or ADVANTIO™ MRI pacemaker with FINELINE™ II Sterox or FINELINE™ II Sterox EZ endocardial pacing lead(s)) when used in the Magnetic Resonance Imaging environment under the labeled Conditions of Use.

DETAILED DESCRIPTION:
Objective of the INFINITE MRI Study is to collect data on the ImageReady MR Conditional Pacing System in subjects undergoing a magnetic resonance scan (MRI).

The ImageReady system has CE mark and enrolled patients will undergo MRI scan under the labeled Conditions of Use. Subjects considered eligible for this studty are already implanted with the system according to standard medical guidelines for PM implantation.

The study is aimed at providing confirmatory data of no impact of MRI on device function, lead parameters and patient conditions. The study will collect standard device measurement through device interrogation pre- and post- MRI scan. MRI scan in this study is a non-clinically indicated procedure and is not planned for diagnostic purposes.

Data from this study will be used to support the evidence of clinical performance of the ImageReady™ MR Conditional Pacing System following a MRI scan when used under the labeled Conditions of Use, and may be used to support regulatory submissions for the approval of the system where requested.

The study has no primary endpoint and is not hypothesis driven.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, or above legal age and willing and capable of giving informed consent specific to national law;
* Patients already implanted with the ImageReady™ MR Conditional Pacing System, single or dual chamber, including INGENIO™ MRI or ADVANTIO™ MRI pulse generators with FINELINE™ II Sterox or FINELINE II Sterox EZ endocardial lead(s), or accessories (see Table 5.1-1) according to standard medical guidelines for pacemaker implantation;
* Willing and capable of participation to the procedures indicated in the protocol.

Exclusion Criteria:

* Patients implanted with pulse generator location outside of left or right pectoral regions;
* Patients implanted with other cardiac-related implanted devices or accessories other than the ImageReadyTM MR Conditional Pacing System;
* Abandoned leads or PGs;
* Evidence of a fractured lead or compromised PG-lead system integrity;
* Low life expectancy (< 1 year);
* Severe comorbidities that, according to clinical judgment, pose patient at risk to undergo MRI;
* Pregnant women or women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients implanted with a ImageReady pacemakers according to standard medical guidelines in the investigational site or referral centers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - ISALA Klinieken, Zwolle

RESULTS

PARTICIPANT FLOW:
Recruitment Details: INFINITE MRI study started subject enrollment on 17 June 2013.Las subject was enrolled on 2 October 2013 and last subject follow up concluded on 17 January 2014. Study database was closed on 28 February 2014.
Period: Overall Study
Arm/Group | ImageReady Pacemaker
Started | 20
Completed | 17
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | ImageReady Pacemaker
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of MRI Related Patient Adverse Events and/or Adverse Device Effects During MRI Visit
Description: The study is aimed at providing confirmatory data of no impact of MRI on device function and patient conditions.
  Confirmation of no MRI related patient adverse events and/or adverse device effects during MRI visit are assessed as follows:
  1. no episodes of asystole,
  2. no occurrence of sustained ventricular arrhythmias in the bore,
  3. no loss of capture due to rise in pacing threshold.
Time Frame: one month
Measure: Number; unit: number of MRI related patient adverse ev
Arm/Group | ImageReady Pacemaker
Number analyzed (Participants) | 17
number of MRI related patient adverse ev | 0

ADVERSE EVENTS:
Arm/Group | ImageReady Pacemaker
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ImageReady Pacemaker (N=20)
atrial fibrillation (Cardiac disorders) | 2 (3)
coronary intervention (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ImageReady Pacemaker (N=20)
paroxisma atrial fibrillation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No